CLINICAL TRIAL: NCT05618080
Title: GRASP-01-003: Trial Readiness and Endpoint Assessment in LGMD R1
Brief Title: LGMD R1 Natural History Study
Acronym: GRASP-01-003
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Nationwide Children's Hospital (Other); Washington University School of Medicine (Other); University of Iowa (Other); University of Florida (Other); University of Minnesota (Other); Newcastle University (Other); University of Kansas Medical Center (Other); University of Colorado, Denver (Other); Indiana CHC (Community Health Clinic) (Unknown); University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HM20025359; Limb-Girdle Muscular Dystrophy (Other: Virginia Commonwealth University); GRASP-R1 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Calpain-3 Deficiency Limb Girdle Muscular Dystrophy Type 2A; Limb Girdle Muscular Dystrophy; Limb Girdle Muscular Dystrophy Type R1; LGMD2A
Keywords: LGMD; Limb Girdle Muscular Dystrophy; LGMD R1; LGMD2A; CAPN3
MeSH Terms: conditions — Limb-girdle muscular dystrophy type 2A; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be taken for biomarker development and retained for future research. No clinical diagnosis will be given to patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGMD Type R1/LGMD2A/CAPN3: No intervention will be administered.

SUMMARY:
This is a 24-month, observational study of 100 participants with Limb Girdle Muscular Dystrophy type R1, also known as CAPN3.

DETAILED DESCRIPTION:
Limb girdle muscular dystrophies (LGMD) are a group of over 30 heterogenous genetic disorders which have in common a pattern of weakness affecting proximal muscles of the shoulders and hips. LGMD type R1 (LGMDR1; also LGMD2A) is due to loss of function of the muscle structural gene calpain 3 (CAPN3) and causes progressive weakness and muscle wasting, which can lead to loss of ambulation or the ability to maintain a job. LGMDR1 is one of the most common LGMDs in the United States and has no FDA approved therapies but is amenable to gene replacement strategies, regenerative medicine approaches, or myostatin based approaches. There have been rapid advances in gene delivery therapies for Duchenne Muscular Dystrophy and for LGMDR4 that have set the stage for targeted therapeutic development for all LGMDs, and LGMDR1 in particular is at a crossroads: the pace of therapeutic development has outstripped the efforts at clinical trial preparedness.

There is a need for a more rigorous natural history study to assist in the design of clinical trials; in particular, identifying biomarkers for early phase development and clinical outcome assessments (COAs) for drug approval studies.

This study will enroll 100 subjects across participating sites in the GRASP-LGMD Research Consortium. No treatment will be administered as part of this study. A subset of 80 patients will undergo MR scans at selected imaging sites. Study visits will occur at Baseline Day 1, Baseline Day 2, Month 12, and Month 24.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12-50 at enrollment
2. Clinically affected (defined as weakness on bedside evaluation in a pattern consistent with LGMDR1)
3. Genetic confirmation of LGMDR1 (presence of homozygous or compound heterozygous pathogenic mutations in CAPN3).
4. Must be able to provide written informed consent and be willing and able to comply with all study requirements. Note: Adult participants must be able to provide consent themselves. Legally authorized representatives are not permitted to consent on behalf of adult participants.

Exclusion Criteria:

1. Have contraindications to MRI or MRS (e.g., non-MR compatible implanted medical devices or severe claustrophobia)
2. Non-ambulatory as defined by those who are not able to walk 10 meters without assistive devices (ankle foot orthotics excluded)
3. Positive pregnancy test at any timepoint during the trial
4. Have dominantly inherited CAPN3 mutations (LGMDD4)
5. Any other illness that would interfere with the ability to undergo safe testing or would interfere with interpretation of the results in the opinion of the site investigator.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes ambulatory individuals aged 12-50 at enrollment who are clinically affected by and have genetic confirmation of LGMDR1.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Validate the NSAD as a clinical outcome assessment in LGMD R1 | Baseline to 24 months
  The North Star Assessment for Dysferlinopathy (NSAD) is a functional scale specifically designed to measure motor performance in individuals with LGMD. It consists of 29 items that are considered clinically relevant items from the North Star Ambulatory Assessment and the Motor Function Measure 20 with a maximum score of 54 and higher scores indicate higher functional abilities.

SECONDARY OUTCOMES:
Validate muscle fat fraction as a biomarker | Baseline to 12 months
  Quantitative muscle MRI (qMR) of the upper and lower leg muscles will be performed and muscle fat fraction will be measured.

OTHER OUTCOMES:
Change in mobility (100-meter walk) | Baseline to 24 months
  Mobility will be measured using the 100 Meter Timed Test (100m) in which the participant is asked to complete 2 laps around 2 cones set 25 meters apart as quickly as safely possible, running if able, and the time in seconds is recorded.
Change in Forced vital capacity (FVC) | Baseline to 24 months
  Volume of air forcefully exhaled will be measured using Spirometry performed in sitting and supine positions using standardized equipment
Change in Forced expiratory volume (FEV1) | Baseline to 24 months
  Volume of air forcefully exhaled in one second will be measured using Spirometry performed in a sitting position using standardized equipment
Change in upper limb function characteristics (PUL) | Baseline to 24 months
  The Performance of Upper Limb 2.0 (PUL) scale measures the progression of weakness and natural history of functional decline in Duchenne muscular dystrophy. There are 22 scored items; a score of 42 indicates the highest level of independent function and 0 the lowest.
Change in Timed Up-And-Go (TUG) | Baseline to 24 months
  Time to stand from a chair, walk 3 meters, and return to seated will be recorded. The test will be repeated three times at applicable visits.
Change in 4 Stair Climb | Baseline to 24 months
  Time to ascend 4 steps as quickly and safely as possible, using handrails if needed, will be assessed.
Change in Handheld Dynamometry and Pinch Grip | Baseline to 24 months
  Maximum hand, pinch, and grip strength will be assessed using a myometer. The participant will be asked to squeeze a handheld tool.
Change in self-reported social, mental, and physical health (PROMIS-57) | Baseline to 24 months
  PROMIS is a set of patient-reported measures developed by the NIH. The social health set of questions evaluates general social health by assessing ability to participate in social roles and activities, companionship, satisfaction with social roles and activities, social isolation, and social support.
  The mental health set evaluates general mental health by assessing anxiety, depression, alcohol use, anger, cognitive function, life satisfaction, meaning and purpose, positive affect, psychosocial illness impact, self-efficacy for managing chronic conditions, smoking, and substance use.
  The physical health set evaluates general physical health by assessing fatigue, pain intensity, pain interference, physical function, sleep disturbance, dyspnea, gastrointestinal symptoms, itch, pain behavior, pain quality, sexual function, and sleep related impairment.
Change in activity limitations (ACTLIVLIM) | Baseline to 24 months
  ACTIVLIM is a patient-reported measure of activity limitations for individuals with upper and/or lower limb impairments, which measures the ability to perform daily activities.
Change in overall health (Domain Delta) | Baseline to 24 months
  Domain Delta Questionnaire is a patient reported measure that assesses overall health over the previous 12 months.
Change in overall health-related quality of life (LGMD-HI) | Baseline to 24 months
  The LGMD Health Index is a disease-specific, patient reported measure that assesses overall health-related quality of life in LGMD.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (12):
- United States (10):
  - University of California, Irvine, Orange, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - The Community Health Clinic, Inc., Shipshewana, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Department of Neurology, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
- Leiden University Medical Center, Leiden, Netherlands
- Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated and deidentified data will be shared with qualified investigators upon majority approval of the LGMD investigators

REFERENCES:
- [Background] van de Velde NM, Hooijmans MT, Sardjoe Mishre ASD, Keene KR, Koeks Z, Veeger TTJ, Alleman I, van Zwet EW, Beenakker JM, Verschuuren JJGM, Kan HE, Niks EH. Selection Approach to Identify the Optimal Biomarker Using Quantitative Muscle MRI and Functional Assessments in Becker Muscular Dystrophy. Neurology. 2021 Aug 3;97(5):e513-e522. doi: 10.1212/WNL.0000000000012233. Epub 2021 Jun 23. PMID 34162720
- [Background] Deenen JC, Horlings CG, Verschuuren JJ, Verbeek AL, van Engelen BG. The Epidemiology of Neuromuscular Disorders: A Comprehensive Overview of the Literature. J Neuromuscul Dis. 2015;2(1):73-85. PMID 28198707
- [Background] Moore SA, Shilling CJ, Westra S, Wall C, Wicklund MP, Stolle C, Brown CA, Michele DE, Piccolo F, Winder TL, Stence A, Barresi R, King N, King W, Florence J, Campbell KP, Fenichel GM, Stedman HH, Kissel JT, Griggs RC, Pandya S, Mathews KD, Pestronk A, Serrano C, Darvish D, Mendell JR. Limb-girdle muscular dystrophy in the United States. J Neuropathol Exp Neurol. 2006 Oct;65(10):995-1003. doi: 10.1097/01.jnen.0000235854.77716.6c. PMID 17021404
- [Background] Nallamilli BRR, Chakravorty S, Kesari A, Tanner A, Ankala A, Schneider T, da Silva C, Beadling R, Alexander JJ, Askree SH, Whitt Z, Bean L, Collins C, Khadilkar S, Gaitonde P, Dastur R, Wicklund M, Mozaffar T, Harms M, Rufibach L, Mittal P, Hegde M. Genetic landscape and novel disease mechanisms from a large LGMD cohort of 4656 patients. Ann Clin Transl Neurol. 2018 Dec 1;5(12):1574-1587. doi: 10.1002/acn3.649. eCollection 2018 Dec. PMID 30564623
- [Background] Arrigoni F, De Luca A, Velardo D, Magri F, Gandossini S, Russo A, Froeling M, Bertoldo A, Leemans A, Bresolin N, D'angelo G. Multiparametric quantitative MRI assessment of thigh muscles in limb-girdle muscular dystrophy 2A and 2B. Muscle Nerve. 2018 Oct;58(4):550-558. doi: 10.1002/mus.26189. Epub 2018 Aug 22. PMID 30028523
- [Background] Barp A, Laforet P, Bello L, Tasca G, Vissing J, Monforte M, Ricci E, Choumert A, Stojkovic T, Malfatti E, Pegoraro E, Semplicini C, Stramare R, Scheidegger O, Haberlova J, Straub V, Marini-Bettolo C, Lokken N, Diaz-Manera J, Urtizberea JA, Mercuri E, Kyncl M, Walter MC, Carlier RY. European muscle MRI study in limb girdle muscular dystrophy type R1/2A (LGMDR1/LGMD2A). J Neurol. 2020 Jan;267(1):45-56. doi: 10.1007/s00415-019-09539-y. Epub 2019 Sep 25. PMID 31555977
- [Background] Feng X, Luo S, Li J, Yue D, Xi J, Zhu W, Gao X, Guan X, Lu J, Liang Z, Zhao C. Fatty infiltration evaluation and selective pattern characterization of lower limbs in limb-girdle muscular dystrophy type 2A by muscle magnetic resonance imaging. Muscle Nerve. 2018 Oct;58(4):536-541. doi: 10.1002/mus.26169. Epub 2018 Sep 3. PMID 29797799
- [Background] Fischer D, Walter MC, Kesper K, Petersen JA, Aurino S, Nigro V, Kubisch C, Meindl T, Lochmuller H, Wilhelm K, Urbach H, Schroder R. Diagnostic value of muscle MRI in differentiating LGMD2I from other LGMDs. J Neurol. 2005 May;252(5):538-47. doi: 10.1007/s00415-005-0684-4. Epub 2005 Feb 23. PMID 15726252
- [Background] Jaka O, Azpitarte M, Paisan-Ruiz C, Zulaika M, Casas-Fraile L, Sanz R, Trevisiol N, Levy N, Bartoli M, Krahn M, Lopez de Munain A, Saenz A. Entire CAPN3 gene deletion in a patient with limb-girdle muscular dystrophy type 2A. Muscle Nerve. 2014 Sep;50(3):448-53. doi: 10.1002/mus.24263. Epub 2014 Aug 5. PMID 24715573
- [Background] Mercuri E, Bushby K, Ricci E, Birchall D, Pane M, Kinali M, Allsop J, Nigro V, Saenz A, Nascimbeni A, Fulizio L, Angelini C, Muntoni F. Muscle MRI findings in patients with limb girdle muscular dystrophy with calpain 3 deficiency (LGMD2A) and early contractures. Neuromuscul Disord. 2005 Feb;15(2):164-71. doi: 10.1016/j.nmd.2004.10.008. Epub 2004 Nov 26. PMID 15694138
- [Background] Willis TA, Hollingsworth KG, Coombs A, Sveen ML, Andersen S, Stojkovic T, Eagle M, Mayhew A, de Sousa PL, Dewar L, Morrow JM, Sinclair CD, Thornton JS, Bushby K, Lochmuller H, Hanna MG, Hogrel JY, Carlier PG, Vissing J, Straub V. Quantitative magnetic resonance imaging in limb-girdle muscular dystrophy 2I: a multinational cross-sectional study. PLoS One. 2014 Feb 28;9(2):e90377. doi: 10.1371/journal.pone.0090377. eCollection 2014. PMID 24587344
- [Background] Reyngoudt H, Marty B, Boisserie JM, Le Louer J, Koumako C, Baudin PY, Wong B, Stojkovic T, Behin A, Gidaro T, Allenbach Y, Benveniste O, Servais L, Carlier PG. Global versus individual muscle segmentation to assess quantitative MRI-based fat fraction changes in neuromuscular diseases. Eur Radiol. 2021 Jun;31(6):4264-4276. doi: 10.1007/s00330-020-07487-0. Epub 2020 Nov 21. PMID 33219846
- [Background] Barnard AM, Willcocks RJ, Finanger EL, Daniels MJ, Triplett WT, Rooney WD, Lott DJ, Forbes SC, Wang DJ, Senesac CR, Harrington AT, Finkel RS, Russman BS, Byrne BJ, Tennekoon GI, Walter GA, Sweeney HL, Vandenborne K. Skeletal muscle magnetic resonance biomarkers correlate with function and sentinel events in Duchenne muscular dystrophy. PLoS One. 2018 Mar 19;13(3):e0194283. doi: 10.1371/journal.pone.0194283. eCollection 2018. PMID 29554116
- [Background] Willcocks RJ, Arpan IA, Forbes SC, Lott DJ, Senesac CR, Senesac E, Deol J, Triplett WT, Baligand C, Daniels MJ, Sweeney HL, Walter GA, Vandenborne K. Longitudinal measurements of MRI-T2 in boys with Duchenne muscular dystrophy: effects of age and disease progression. Neuromuscul Disord. 2014 May;24(5):393-401. doi: 10.1016/j.nmd.2013.12.012. Epub 2014 Jan 11. PMID 24491484
- [Background] Burakiewicz J, Sinclair CDJ, Fischer D, Walter GA, Kan HE, Hollingsworth KG. Quantifying fat replacement of muscle by quantitative MRI in muscular dystrophy. J Neurol. 2017 Oct;264(10):2053-2067. doi: 10.1007/s00415-017-8547-3. Epub 2017 Jul 1. PMID 28669118
- [Background] Willcocks RJ, Rooney WD, Triplett WT, Forbes SC, Lott DJ, Senesac CR, Daniels MJ, Wang DJ, Harrington AT, Tennekoon GI, Russman BS, Finanger EL, Byrne BJ, Finkel RS, Walter GA, Sweeney HL, Vandenborne K. Multicenter prospective longitudinal study of magnetic resonance biomarkers in a large duchenne muscular dystrophy cohort. Ann Neurol. 2016 Apr;79(4):535-47. doi: 10.1002/ana.24599. Epub 2016 Feb 19. PMID 26891991
- [Background] Comi GP, Niks EH, Cinnante CM, Kan HE, Vandenborne K, Willcocks RJ, Velardo D, Ripolone M, van Benthem JJ, van de Velde NM, Nava S, Ambrosoli L, Cazzaniga S, Bettica PU. Characterization of patients with Becker muscular dystrophy by histology, magnetic resonance imaging, function, and strength assessments. Muscle Nerve. 2022 Mar;65(3):326-333. doi: 10.1002/mus.27475. Epub 2021 Dec 30. PMID 34918368
- [Background] Batra A, Lott DJ, Willcocks R, Forbes SC, Triplett W, Dastgir J, Yun P, Reghan Foley A, Bonnemann CG, Vandenborne K, Walter GA. Lower Extremity Muscle Involvement in the Intermediate and Bethlem Myopathy Forms of COL6-Related Dystrophy and Duchenne Muscular Dystrophy: A Cross-Sectional Study. J Neuromuscul Dis. 2020;7(4):407-417. doi: 10.3233/JND-190457. PMID 32538860
- [Background] Hung M, Clegg DO, Greene T, Saltzman CL. Evaluation of the PROMIS physical function item bank in orthopaedic patients. J Orthop Res. 2011 Jun;29(6):947-53. doi: 10.1002/jor.21308. Epub 2011 Mar 15. PMID 21437962
- [Background] Hung M, Baumhauer JF, Brodsky JW, Cheng C, Ellis SJ, Franklin JD, Hon SD, Ishikawa SN, Latt LD, Phisitkul P, Saltzman CL, SooHoo NF, Hunt KJ; Orthopaedic Foot & Ankle Outcomes Research (OFAR) of the American Orthopaedic Foot & Ankle Society (AOFAS). Psychometric Comparison of the PROMIS Physical Function CAT With the FAAM and FFI for Measuring Patient-Reported Outcomes. Foot Ankle Int. 2014 Jun;35(6):592-599. doi: 10.1177/1071100714528492. PMID 24677217
- [Background] Christensen KB, Makransky G, Horton M. Critical Values for Yen's Q3: Identification of Local Dependence in the Rasch Model Using Residual Correlations. Appl Psychol Meas. 2017 May;41(3):178-194. doi: 10.1177/0146621616677520. Epub 2016 Nov 16. PMID 29881087
- [Background] Khadka J, Pesudovs K, McAlinden C, Vogel M, Kernt M, Hirneiss C. Reengineering the glaucoma quality of life-15 questionnaire with rasch analysis. Invest Ophthalmol Vis Sci. 2011 Sep 1;52(9):6971-7. doi: 10.1167/iovs.11-7423. PMID 21810983
- [Background] Hung M, Voss MW, Bounsanga J, Gu Y, Granger EK, Tashjian RZ. Psychometrics of the Patient-Reported Outcomes Measurement Information System Physical Function instrument administered by computerized adaptive testing and the Disabilities of Arm, Shoulder and Hand in the orthopedic elbow patient population. J Shoulder Elbow Surg. 2018 Mar;27(3):515-522. doi: 10.1016/j.jse.2017.10.015. Epub 2018 Jan 9. PMID 29325704